CLINICAL TRIAL: NCT05554068
Title: Phase II, Non-randomized, Open-label Study to Assess the Immunogenicity and Clinical Efficacy of the Recombinant Zoster Vaccine for Recipients of an Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Immunogenicity of Zoster Vaccine in Allogeneic Hematopoietic Stem Cell Transplant Recipients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Hagen, Patrick A, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215468
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Shingles
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shingrix (Experimental): Patients 1-3 years post transplant will receive the Shingrix vaccine in standard dosing and schedule.
  Interventions: Drug: Shingrix

INTERVENTIONS:
Drug: Shingrix — Shingrix vaccine will be given to all eligible patients at one to three year post allogeneic stem cell transplantation.

SUMMARY:
This is a phase II study that will examine the immunogenicity of the Shingrix vaccine in patients following an allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Cell mediated immunity is severely compromised after an allogeneic stem cell transplantation. This results in an increased risk of zoster with its associated morbidity and mortality. Patients typically receive prophylactic antivirals for 1 year after AlloSCT which reduces the incidence of zoster during this period. Unfortunately, after completing prophylaxis, patients continue to be at a significantly increased risk of zoster with an incidence rate of up to 29% at 3-years post transplant. The recombinant zoster vaccine provides immunogenicity and has shown clinical efficacy in preventing zoster in patients who have received an autologous transplant.

Furthermore, it has been shown to be safe in patients who had received an allogeneic transplant in a retrospective study although immunogenicity seemed to be decreased in this cohort. Due to the paucity of data in allogeneic recipients, we propose a prospective, non-randomized study to evaluate the immunogenicity and clinical efficacy of the recombinant zoster vaccine in recipients of allogeneic stem cell transplantation. As a secondary endpoint, we will compare our results to historical data of immunogenicity and clinical effectiveness of the vaccine in autologous transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ≥ 12 months and ≤ 36 months post-AlloSCT
* Donor sources: matched related, matched unrelated, cord blood
* Any malignant hematological disease including acute leukemia, myelodysplastic syndrome, non-Hodgkin's lymphoma, Hodgkin's lymphoma, chronic lymphocytic leukemia, chronic myeloid leukemia, multiple myeloma, and myeloproliferative disorders.
* Any conditioning regimen
* Any planned immunosuppressive prophylactic regimen
* Patients with chronic graft-versus-host disease on stable immunosuppression
* Ability to understand and the willingness to sign a written informed consent.
* Negative pregnancy test in female patients of childbearing potential

Exclusion Criteria:

* Patients who had zoster after an allogeneic transplant and prior to enrollment
* Patients who are currently pregnant
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the recombinant zoster vaccine, Shingrix, or other agents used in study.
* Patients who have had a relapse of their primary hematological disease
* Previous allogeneic stem cell transplantation
* Acute disease at the time of vaccination
* Thrombocytopenia that in the judgment of the investigator would make intramuscular injection unsafe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Cell mediated and humoral immune response | Measured one month following eh last dose of vaccine received

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No